CLINICAL TRIAL: NCT06783998
Title: Evaluation of Respiratory Muscle Sarcopenia in Obstructive Sleep Apnea Syndrome
Acronym: RMS-OSAS
Status: Enrolling by invitation | Type: Observational
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Nurel Ertürk, Assist. Prof. PT. PhD Nurel Ertürk, Tarsus University
Other Study IDs: 2025/01
Record Dates: First submitted 2025-01-06; First posted 2025-01-20 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea (OSAS)
Keywords: Obstruktive sleep apnea; sarcopenia; respiratory muscle
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OSAS: Turkish-speaking patients diagnosed with normal-mild-moderate-severe OSAS, aged 18 and over, will be included.

SUMMARY:
OSAS is a disease characterized by repeated interruptions and restarts of breathing during sleep. Respiratory muscle sarcopenia is a condition in which the muscle strength of the diaphragm and other respiratory auxiliary muscles decreases, resulting in a decrease in breathing effort. Decreased respiratory effort is an important indicator of OSAS. Age, presence of chronic disease, and obesity increase the presence and severity of respiratory sarcopenia. If OSAS is left untreated, it leads to cardiovascular diseases, dementia, Alzheimer's and even death in early adulthood. In recent years, studies have shown that continuous positive airway pressure (CPAP), as well as healthy behavior development, preventive health and exercise measures, are important in the management of these diseases. There is no research in the literature on the evaluation of respiratory muscle sarcopenia in OSAS patients.

This study aims to evaluate respiratory muscle sarcopenia in OSAS based on a concrete value reflecting respiratory muscle strength and/or volume.

DETAILED DESCRIPTION:
In the study, respiratory muscle sarcopenia will be evaluated in OSAS patients. It will be evaluated whether the expiratory pressure value, peek flow meter value and 6-minute walking distance are predictors of respiratory sarcopenia for OSAS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with normal-mild-medium-severe OSAS
* 18 years and above
* Turkish speaking patients will be included.

Exclusion Criteria:

* Pregnancy,

  * Latent autoimmune diabetes,
  * Chronic renal failure,
  * Active or serious infections,
  * Liver failure,
  * Recent major cardiovascular events,
  * Unstable angina, heart failure (NYHA III-IV),
  * Patients with neurological or musculoskeletal disorders that create limitations in walking and performing tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with normal-mild-medium-severe Obstructive Sleep Apnea Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Anthropometric measurement | 1 year
  Waist circumference, hip circumference will be measured, waist-hip ratio will be calculated.
BOdy mass measurement | 1 year
  Body weight,fat-free mass (FFM) and appendicular skeletal muscle mass (ASMM) and skeletal muscle mass expressed in kilograms will be measured by bioelectrical impedance.
Hand Grip strength | 1 year
  Jamar hand dynamometer, which is recommended by the American Association of Hand Therapists (AETD) and has been found to have high validity and reliability in many studies and is therefore considered the gold standard, will be used to measure hand grip strength.
Walking speed | 1 year
  Walking speed will be measured with the 4 Meter Walking Speed Test (4MYHT).
Respiratory muscle strength: | 1 year
  Respiratory muscle strength will be evaluated with a portable, electronic mouth pressure measurement device.
Expiratory flow rate | 1 year
  Peak expiratory flow (PEF), also called peak expiratory flow rate (PEFR) and peak flow measurement, will be measured with a PEFmeter (MSA 100 PEFmeter), a small, hand-held device used to monitor a person's ability to breathe air.
Respiratory function test | 1 year
  To evaluate pulmonary functions(FEV1/FVC ve FEV1 ), it will be measured in a sitting position with a Spirolab III brand spirometer according to ATS/European Respiratory Society (ERS) criteria.

SECONDARY OUTCOMES:
Functional capacity | 1 year
  Functional exercise capacity will be evaluated with the 6-minute walk test (6MWT)

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No